CLINICAL TRIAL: NCT00108953
Title: A Randomized Controlled Study of BAY43-9006 in Combination With Doxorubicin Versus Doxorubicin in Patients With Advanced Hepatocellular Carcinoma.
Brief Title: A Research Study to Treat Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11546; 2004-001770-40 (EudraCT Number)
Record Dates: First submitted 2005-04-21; First posted 2005-04-22 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Cancer; Liver Cancer; Hepatocellular carcinoma; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Liver Neoplasms | interventions — Sorafenib; Doxorubicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib + Doxorubicin (Experimental): "Sorafenib + Doxorubicin" -- combination therapy: Sorafenib (Nexavar, BAY43-9006) 200 mg tablets by mouth (orally) twice daily + doxorubicin 60 mg/m2 intravenous infusion every 21 days for 6 cycles (18 weeks)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006) plus Doxorubicin
- Placebo + Doxorubicin (Active Comparator): "Placebo + Doxorubicin" -- monotherapy: Sorafenib (Nexavar, BAY43-9006) matching placebo tablets by mouth (orally) twice daily + doxorubicin 60 mg/m2 intravenous infusion every 21 days for 6 cycles (18 weeks)
  Interventions: Drug: Doxorubicin/Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) plus Doxorubicin — Multi kinase inhibitor plus Chemotherapy
  Arms: Sorafenib + Doxorubicin
Drug: Doxorubicin/Placebo — Chemotherapy plus Placebo
  Arms: Placebo + Doxorubicin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of doxorubicin plus sorafenib versus doxorubicin plus placebo in patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
In addition to the key secondary outcome parameters the following parameters will be assessed in an exploratory manner: relative time to progression (TTP), time to symptomatic progression (TTSP), response rate (RR) and overall survival between the 2 study populations.

The possible and potential predictive assays of clinical benefit through an assessment of the correlation between the defined baseline characteristics and key clinical endpoints.

The safety and tolerability will be assessed in the adverse event section. Doxorubicin pharmacokinetics in HCC patients treated with sorafenib versus placebo will be compared and the pharmacokinetic data will be correlated with doxorubicin-related adverse events (i.e., cardiotoxicity).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a life expectancy of at least 12 weeks
* Patients with advanced HCC (unresectable, and/or metastatic) which has been histologically or cytologically documented
* Patients must have at least one tumor lesion that meets both of the following criteria:

  * can be accurately measured in at least one dimension according to Response Evaluation Criteria in Solid Tumors (RECIST)
  * has not been previously treated with local therapy
* Patients who have received local therapy except chemoembolization, such as surgery, radiation therapy, hepatic arterial embolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation are eligible, provided that they either have a target lesion which has not been subjected to local therapy and/or the target lesion(s) within the field of the local therapy has shown an increase of 25% in the size. Local therapy must be completed at least 4 weeks prior to the baseline scan
* Patients who have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted
* History of cardiac disease
* Serious myocardial dysfunction
* Active, clinically serious infections
* Known history of Human Immunodeficiency Virus (HIV) infection
* Known Central Nervous System (CNS) tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- United States (14):
  - Birmingham, Alabama
  - Beverly Hills, California
  - Orange, California
  - Palo Alto, California
  - San Francisco, California
  - Sylmar, California
  - Miami, Florida
  - Lafayette, Louisiana
  - Minneapolis, Minnesota
  - Hackensack, New Jersey
  - New York, New York
  - Rochester, New York
  - Nashville, Tennessee
  - Seattle, Washington
- Argentina (3):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Neuquén, Neuquén Province
  - Buenos Aires
- Toronto, Ontario, Canada
- Hong Kong, Hong Kong, Hong Kong
- Russia (3):
  - Kazan'
  - Kirov
  - Krasnodar
- United Kingdom (5):
  - Maidstone, Kent
  - London, London
  - Manchester, Manchester
  - Bebington, Merseyside
  - Birmingham, West Midlands

REFERENCES:
- [Result] Abou-Alfa GK, Schwartz L, Ricci S, Amadori D, Santoro A, Figer A, De Greve J, Douillard JY, Lathia C, Schwartz B, Taylor I, Moscovici M, Saltz LB. Phase II study of sorafenib in patients with advanced hepatocellular carcinoma. J Clin Oncol. 2006 Sep 10;24(26):4293-300. doi: 10.1200/JCO.2005.01.3441. Epub 2006 Aug 14. PMID 16908937
- [Result] Abou-Alfa GK, Johnson P, Knox JJ, Capanu M, Davidenko I, Lacava J, Leung T, Gansukh B, Saltz LB. Doxorubicin plus sorafenib vs doxorubicin alone in patients with advanced hepatocellular carcinoma: a randomized trial. JAMA. 2010 Nov 17;304(19):2154-60. doi: 10.1001/jama.2010.1672. PMID 21081728
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started on 13 Apr 2005 and the last study contact occurred on 11 Apr 2008. The study was conducted at 25 active centers in 6 countries (Argentina, Canada, Hong Kong, Russia, United Kingdom, and United States.)
Pre-assignment Details: 140 patients were screened, with 44 screen failures. The intent-to-treat (ITT) population (primary efficacy analysis) includes all randomized patients (96). The Safety population includes all patients who received at least 1 dose of study drug (95). The study consists of 2 periods: treatment period (not fixed but ended by any event) and follow-up.
Period: Treatment Period
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Started | 47 (ITT population) | 49 (ITT population)
Completed | 47 (No patient under study medication anymore) | 49 (No patient under study medication anymore)
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Started | 40 (40 out of 47 patients were followed after end of double blind treatment) | 45 (45 out of 49 patients were followed after end of double blind treatment)
Completed | 11 | 12
Not Completed | 29 | 33
Not completed — Death | 18 | 26
Not completed — Lost to Follow-up | 1 | 1
Not completed — Study terminated by sponsor | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Continuous [Median (Full Range); unit: years]
  Median (Full Range) | 66 [38 to 82] | 65 [38 to 81] | 65 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 31 | 42 | 73
Child Pugh Status [Number; unit: participants] — The Child-Pugh score is used to classify the stages of liver cirrhosis, based on clinical diagnosis and laboratory tests. Assessment of good operative risk (A) if 5 or 6 points, moderate risk (B) if 7 to 9 points, and poor operative risk (C) if 10 to 15 points. A "C" classification forecasts a survival of less than 12 months.
  participants
    5 (Child-Pugh A) | 30 | 28 | 58
    6 (Child-Pugh A) | 17 | 19 | 36
    7 (Child-Pugh B) | 0 | 2 | 2
    >7 | 0 | 0 | 0
Eastern Cooperative Group performance status (ECOG PS) at study entry [Number; unit: participants] — ECOG PS is a rating of daily living abilities, from 0 to 5. 0=Fully active without restriction. 1= Restricted in physically strenuous activity; 2= Ambulatory, capable of all selfcare; 3= Capable of limited selfcare; 4= Completely disabled; 5= Dead.
  participants
    Grade 0 | 22 | 16 | 38
    Grade 1 | 18 | 25 | 43
    Grade 2 | 4 | 3 | 7
    Grade 3 | 0 | 1 | 1
    missing | 3 | 4 | 7
Tumor burden: Extrahepatic spread [Number; unit: participants] — Tumor spread outside the liver, which describes an aggressive and advanced tumor pattern.
  participants
    yes | 24 | 32 | 56
    no | 23 | 17 | 40
Tumor burden: Macroscopic vascular invasion [Number; unit: participants] — Tumor spread into the blood vessels as determined through radiological assessment (e.g., x-ray, imaging), which describes an aggressive and advanced tumor pattern.
  participants
    yes | 13 | 16 | 29
    no | 33 | 32 | 65
    missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from randomization to radiological disease progression by independent assessment.
Time Frame: from date of randomization of the first patient until 3 years later
Population: The intent-to-treat (ITT) population, primary population for efficacy analysis, includes all randomized patients.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
days | 263 [146 to 384] | 147 [66 to 244]
Statistical Analysis 1: Comparison: Sorafenib + Doxorubicin vs Placebo + Doxorubicin; The comparison between the 2 groups is done using the log rank test stratified by tumor burden. The null hypothesis is: TTP is the same in both treatment groups; Test type: Superiority or Other; p = 0.016, Log Rank; Hazard Ratio, log = 0.6, 95% CI [0.33 to 0.95] — Hazard ratio: nexavar+doxorubicin over placebo+doxorubicin

2. Secondary Outcome: Overall Survival
Description: The time from date of randomization to date of death
Time Frame: from date of randomization of the first patient until 3 years later
Population: The ITT population, primary population for efficacy analysis, includes all randomized patients. The table below gives the lower and upper limit of the confidence interval; 999999999 = not estimable.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
days | 418 [317 to 999999999] | 199 [148 to 302]
Statistical Analysis 1: Comparison: Sorafenib + Doxorubicin vs Placebo + Doxorubicin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.007, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI [0.37 to 0.74] — Hazard ratio: nexavar+doxorubicin over placebo+doxorubicin

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from the date of randomization to the date of the first documented radiological progression (as defined per independent central radiological assessment) or death, whichever occurs first
Time Frame: from date of randomization of the first patient until 3 years later
Population: The ITT population, primary population for efficacy analysis, includes all randomized patients.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Sorafenib + Doxorubicin: "Sorafenib + Doxorubicin" -- combination therapy: Sorafenib (Nexavar, BAY 43-9006) 200 mg tablets by mouth (orally) twice daily + doxorubicin 60 mg/m2 intravenous infusion every 21 days for 6 cycles (18 weeks)
- Placebo + Doxorubicin: "Placebo + Doxorubicin" -- monotherapy: Sorafenib (Nexavar, BAY 43-9006) matching placebo tablets by mouth (orally) twice daily + doxorubicin 60 mg/m2 intravenous infusion every 21 days for 6 cycles (18 weeks)
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
days | 242 [140 to 312] | 85 [71 to 172]
Statistical Analysis 1: Comparison: Sorafenib + Doxorubicin vs Placebo + Doxorubicin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.018, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI [0.45 to 0.83] — Hazard ratio: nexavar+doxorubicin over placebo+doxorubicin

4. Secondary Outcome: Percentage of Participants in Each Category of Best Tumor Response
Description: Percentage of participants with complete or partial response (CR or PR) confirmed according to Response Evaluation Criteria in Solid Tumors (RECIST) and achieved during treatment or 30 days after end of treatment. CR: disappearance of all clinical and radiological tumor lesions. PR: at least 30% decrease in sum of the longest diameters of tumor lesions. Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase for progressive disease.
Time Frame: achieved during treatment or within 30 days after termination of active therapy
Population: The ITT population, primary population for efficacy analysis, includes all randomized patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
Percentage of participants
  Complete Response (CR) | 0.0 | 2.0
  Partial Response (PR) | 4.3 | 0.0
  Stable Disease (SD) | 66.0 | 49.0

5. Secondary Outcome: Time to Symptomatic Progression (TTSP)
Description: Time from date of randomization to date of first documented symptomatic progression defined by Functional Assessment of Cancer Therapy Hepatobiliary Symptom Index-8 (FHSI-8) assessment
Time Frame: from date of randomization of the first patient until 3 years later
Population: The ITT population, primary population for efficacy analysis, includes all randomized patients.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
days | 208 [85 to 317] | 152 [110 to 180]
Statistical Analysis 1: Comparison: Sorafenib + Doxorubicin vs Placebo + Doxorubicin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.038, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI [0.40 to 1.05] — Hazard ratio: nexavar+doxorubicin over placebo+doxorubicin

6. Secondary Outcome: Duration of Response
Description: Time from date of first objective response (complete response [CR] or partial response [PR]) to date progression is first documented (as defined per independent central radiological assessment) or death, whichever occurs first
Time Frame: from date of randomization of the first patient until 3 years later
Population: The ITT population, primary population for efficacy analysis, includes all randomized patients.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
days | 199 [97 to 301] | 68 [68 to 68]

7. Secondary Outcome: Time to Response (TTR)
Description: Time from date of randomization to date of first objective response (complete response [CR] or partial response [PR]) is documented and confirmed according to RECIST criteria
Time Frame: from date of randomization until 3 years later at end of study
Population: The ITT population, primary population for efficacy analysis, includes all randomized patients.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
days | 134 [83 to 184] | 40 [40 to 40]

8. Secondary Outcome: Percentage of Participants for Whom Disease Control Was Achieved
Description: Participants with disease control: those who have as best response complete response (CR), partial response (PR) or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase for progressive disease) according to Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: from date of randomization to end of treatment plus 30 days
Population: The ITT population, primary population for efficacy analysis, includes all randomized patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Number analyzed (Participants) | 47 | 49
Percentage of participants | 63.8 | 30.6

ADVERSE EVENTS:
Description: The following abbreviations were used in the Adverse Event section:
  * Common toxicity criteria for adverse events (CTCAE)
  * Absolute neutrophil count (ANC)
  * Alanine aminotransferase (AST)
  * Gastrointestinal (GI)
  * Not otherwise specified (NOS)
  * International normalized ratio (INR)
  * Alanine aminotransferase (ALT)
Arm/Group | Sorafenib + Doxorubicin | Placebo + Doxorubicin
Serious Adverse Events (participants affected / at risk) | 19/47 | 20/48
Other Adverse Events (participants affected / at risk) | 47/47 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Doxorubicin (N=47) | Placebo + Doxorubicin (N=48)
Neutrophils (Blood and lymphatic system disorders) | 2 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1
Supraventricular Arrhythmia, Atrial Fibrillation (Cardiac disorders) | 1 | 1
Supraventricular Arrhythmia, Sinus Tachycardia (Cardiac disorders) | 1 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 2 | 0
Hypotension (Cardiac disorders) | 0 | 1
Death not associated with CTCAE term, Disease Progression NOS (General disorders) | 3 | 10
Fever (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0
Mucositis (Clinical Exam), Oral Cavity (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI, Stomach (Vascular disorders) | 1 | 0
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 1 | 0
Liver Dysfunction (Hepatobiliary disorders) | 1 | 0
Hepathobilary - other (Hepatobiliary disorders) | 0 | 1
Febrile Neutropenia (Infections and infestations) | 1 | 5
Infection with normal ANC, Skin (Cellulitis) (Infections and infestations) | 2 | 0
Infection (Documented Clinically), Blood (Infections and infestations) | 1 | 0
Infection (Documented Clinically), Kidney (Infections and infestations) | 1 | 0
Infection (Documented Clinically), Lung (Pneumonia) (Infections and infestations) | 0 | 1
Infection (Documented Clinically), Skin (Cellulitis) (Infections and infestations) | 1 | 0
Infection with normal ANC, Soft Tissue NOS (Infections and infestations) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Lipase (Metabolism and nutrition disorders) | 1 | 1
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Neurology - other (Nervous system disorders) | 0 | 1
Pain, Back (General disorders) | 2 | 1
Pain, Abdomen NOS (General disorders) | 2 | 1
Pain, Chest/Thorax NOS (General disorders) | 1 | 0
Pain, Liver (General disorders) | 1 | 0
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 | 1
Artery Injury, Visceral (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Doxorubicin (N=47) | Placebo + Doxorubicin (N=48)
Neutrophils (Blood and lymphatic system disorders) | 31 | 29
Hemoglobin (Blood and lymphatic system disorders) | 15 | 15
Leukocytes (Blood and lymphatic system disorders) | 10 | 9
Fatigue (General disorders) | 39 | 32
Insomnia (General disorders) | 13 | 8
Nausea (Gastrointestinal disorders) | 27 | 27
Constipation (Gastrointestinal disorders) | 21 | 21
Anorexia (Gastrointestinal disorders) | 24 | 14
Diarrhea (Gastrointestinal disorders) | 25 | 12
Mucositis (Functional/Symptomatic), Oral Cavity (Gastrointestinal disorders) | 11 | 14
GI - other (Gastrointestinal disorders) | 13 | 7
Mucositis (Clinical Exam), Oral Cavity (Gastrointestinal disorders) | 10 | 6
Taste Alteration (Gastrointestinal disorders) | 10 | 5
Edema: Limb (Blood and lymphatic system disorders) | 15 | 14
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 15 | 15
AST (Metabolism and nutrition disorders) | 11 | 7
Dizziness (Nervous system disorders) | 10 | 4
Pain, Abdomen NOS (General disorders) | 18 | 15
Pain, Back (General disorders) | 14 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 25
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 18 | 8
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 14 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 10 | 4
Vomiting (Gastrointestinal disorders) | 17 | 10
Rhinits (Immune system disorders) | 4 | 5
Blood Other (Blood and lymphatic system disorders) | 6 | 7
Platelets (Blood and lymphatic system disorders) | 7 | 9
INR (Blood and lymphatic system disorders) | 0 | 3
Supraventricular Arrhythmia, Sinus Tachycardia (Cardiac disorders) | 4 | 0
Hypertension (Cardiac disorders) | 8 | 0
Hypotension (Cardiac disorders) | 0 | 4
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 9 | 0
Fever (General disorders) | 4 | 4
Weight Loss (General disorders) | 9 | 7
Constitutional Symptoms- Other (General disorders) | 7 | 0
Rigors/Chills (General disorders) | 5 | 0
Sweating (General disorders) | 3 | 4
Ascites (Gastrointestinal disorders) | 4 | 6
Distention (Gastrointestinal disorders) | 5 | 6
Dry Mouth (Gastrointestinal disorders) | 4 | 4
Dysphagia (Gastrointestinal disorders) | 7 | 0
Flatulence (Gastrointestinal disorders) | 3 | 4
Hemorrhoids (Gastrointestinal disorders) | 0 | 3
Heartburn (Gastrointestinal disorders) | 5 | 3
Teeth (Gastrointestinal disorders) | 3 | 0
Hemorrhage, GI, Oral Cavity (Vascular disorders) | 3 | 0
Hemorrhage Pulmonary, Nose (Vascular disorders) | 5 | 3
Liver Dysfunction (Gastrointestinal disorders) | 0 | 3
Infection(Documented Clinically), Oral cavity - gums (Infections and infestations) | 6 | 3
Febrile Neutropenia (Infections and infestations) | 0 | 3
Infection- Other (Infections and infestations) | 3 | 3
Musculoskeletal- Other (Musculoskeletal and connective tissue disorders) | 8 | 4
Alkaline Phosphatase (Metabolism and nutrition disorders) | 5 | 7
ALT (Metabolism and nutrition disorders) | 8 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0
Metabolic/Lab- Other (Metabolism and nutrition disorders) | 3 | 5
Mood Alteration, Anxiety (Nervous system disorders) | 3 | 3
Mood Alteration, Depression (Nervous system disorders) | 4 | 0
Neuropathy: sensory (Nervous system disorders) | 7 | 4
Ocular- Other (Eye disorders) | 4 | 0
Watery Eye (Eye disorders) | 3 | 0
Pain, Chest Wall (General disorders) | 3 | 3
Pain, Extremity-Limb (General disorders) | 3 | 0
Pain, Head/Headache (General disorders) | 9 | 6
Pain, Joint (General disorders) | 9 | 3
Pain, Muscle (General disorders) | 6 | 0
Pain, Other (General disorders) | 5 | 3
Pain, Liver (General disorders) | 6 | 3
Pain, Middle Ear (General disorders) | 3 | 0
Pain, Pain NOS (General disorders) | 3 | 0
Pain, Stomach (General disorders) | 3 | 0
Pain, Throat/Pharynx/Larynx (General disorders) | 3 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pulmonary- Other (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnea(Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 0
Bruising (Skin and subcutaneous tissue disorders) | 6 | 3
Nail changes (Skin and subcutaneous tissue disorders) | 5 | 0
Dermatology- Other (Skin and subcutaneous tissue disorders) | 8 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 3
Flushing (Skin and subcutaneous tissue disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
The study had been prematurely terminated by the sponsor because positive results were obtained in another Nexavar trial (Phase 3 study 100554 NCT00105443). NCI-CTC was translated to MedDRA for SOCs only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution of the Coordinating Investigator (CI) has the right, consistent with academic standards, to publish any proposed publication written by the consultant as part of their services under this agreement. If the sponsor believes that any proposed publication contained any confidential information, the sponsor shall notify the CI, and the CI shall remove such confidential information.